CLINICAL TRIAL: NCT01107158
Title: The Role of Two Nuclear Receptors for Oxysterols as a Molecular Cause of Uterine Dystocia: LXR Alpha and LXR Beta
Brief Title: LXRs, Cholesterol Metabolism and Uterine Dystocia
Status: Terminated | Type: Observational
Why Stopped: Inclusion curve too slow.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2009/KM-01; 2009-A00968-49 (Other: ANSM)
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-11

CONDITIONS: Uterine Inertia; Dystocia
MeSH Terms: conditions — Uterine Inertia; Dystocia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A whole blood sample is taken and DNA extracted using Qiagen kits.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Control group: these patients have mechanical dystocia; cholesterol metabolism factors are a priori not involved.
  Interventions: Biological: Whole blood sampling
- Group 2: These patients have uterine dystocia
  Interventions: Biological: Whole blood sampling

INTERVENTIONS:
Biological: Whole blood sampling — Whole blood sampling for SNP polymorphism analysis

SUMMARY:
Despite the fact that a link between cholesterol and the myometrium has been clearly established, no study investigating aspects of cholesterol metabolism and uterine dystocia currently exists. This study is a pilot study whose aim is to test the hypothesis that an association between uterine dystocia and single-nucleotide polymorphisms (SNPs) in the genes coding for the LXRs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing C-section for a dystocia: 2 to 3 hours of stagnation in labor progress are observed (ie no increasing dilation, and uterine contractions less that 3-5 per 10 minutes) in spite of measures taken to overcome dystocia (oxytocin injection and artificial breaking of waters)
* the child is alive
* the child does not have apriori known malformations that could interfere with a vaginal birth
* foetus in cephalic position
* full term pregnancy (>= 37 weeks of amenorrhea)
* single birth
* patient has signed consent
* patient is affiliated with a social security system

Exclusion Criteria:

* vaginal birth
* programmed C-section
* C-section is chosen because the fetus has a cardia rhythm problem, and there is no stagnation in the labor process
* multiple pregnancy
* the child is in a breech position
* premature birth (<37 weeks amenorrhea)
* in utero fetal death
* fetal malformation known before birth that could interfere with a vaginal birth
* non french-speaking patient (impossible to correctly inform the patient)
* patient under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population represents women undergoing a difficult, stagnating labor due to either physical or uterine dystocia.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2010-04; Primary Completion 2015-09-03 (Actual); Study Completion 2015-09-03 (Actual)

PRIMARY OUTCOMES:
The multi-loci genotype of the target DNA sequence. | Day 1
  The polymorphisms of interest are the following SNPs: rs3758673, rs3758674, rs12221497, rs11039155, rs2279238, rs7120118, rs35463555, rs1052533, rs2248949, rs41432149, rs1405655, rs4802703.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mouzat, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, France

REFERENCES:
- [Result] Mouzat K, Raoul C, Polge A, Kantar J, Camu W, Lumbroso S. Liver X receptors: from cholesterol regulation to neuroprotection-a new barrier against neurodegeneration in amyotrophic lateral sclerosis? Cell Mol Life Sci. 2016 Oct;73(20):3801-8. doi: 10.1007/s00018-016-2330-y. Epub 2016 Aug 10. PMID 27510420